CLINICAL TRIAL: NCT07349680
Title: Ultrasound-Guided Thoracic Paravertebral Block With Steroid and Local Anesthetic for Acute Herpes Zoster: Effects on Pain Control and Prevention of Postherpetic Neuralgia: A Randomized Controlled Trial
Brief Title: Ultrasound-Guided Thoracic Paravertebral Block With Steroid and Local Anesthetic for Acute Herpes Zoster: Effects on Pain Control and Prevention of Postherpetic Neuralgia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marwa mahmoud Abd El Rady, clinical proffessor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20260230004
Record Dates: First submitted 2026-01-14; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Postherpetic Neuralgia
MeSH Terms: conditions — Neuralgia, Postherpetic | interventions — Valacyclovir; Acetaminophen; Gabapentin; Methylprednisolone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard medical therapy for acute thoracic herpes zoster (Other): Participants received standard medical therapy consisting of:
  Valacyclovir 1000 mg orally three times daily for 7 days
  Paracetamol (Acetaminophen) 1 g orally twice daily for 14 days
  Gabapentin starting at 300 mg/day, titrated according to pain intensity and tolerance, up to a maximum of 1800 mg/day
  Interventions: Drug: Valacyclovir + Paracetamol (Acetaminophen) + Gabapentin (standard medical therapy)
- Ultrasound-guided thoracic paravertebral block (TPVB) with local anesthetic + corticosteroid (Active Comparator): Participants received an ultrasound-guided thoracic paravertebral block (TPVB) using an injectate volume of 15 mL, consisting of:
  Bupivacaine 0.25% (local anesthetic)
  Methylprednisolone 40 mg (corticosteroid)
  The block was performed at the thoracic level corresponding to maximal pain/dermatomal involvement, and was repeated every 48 hours for a total of three sessions.
  Interventions: Drug: Valacyclovir + Paracetamol (Acetaminophen) + Gabapentin (standard medical therapy); Procedure: Ultrasound-guided thoracic paravertebral block (TPVB) with bupivacaine 0.25% + methylprednisolone 40 mg

INTERVENTIONS:
Drug: Valacyclovir + Paracetamol (Acetaminophen) + Gabapentin (standard medical therapy) — Participants received standard medical therapy consisting of:
  Valacyclovir 1000 mg orally three times daily for 7 days
  Paracetamol (Acetaminophen) 1 g orally twice daily for 14 days
  Gabapentin starting at 300 mg/day, titrated according to pain intensity and tolerance, up to a maximum of 1800 mg/day
Procedure: Ultrasound-guided thoracic paravertebral block (TPVB) with bupivacaine 0.25% + methylprednisolone 40 mg — Participants received an ultrasound-guided thoracic paravertebral block (TPVB) using an injectate volume of 15 mL, consisting of:
  Bupivacaine 0.25% (local anesthetic)
  Methylprednisolone 40 mg (corticosteroid)
  The block was performed at the thoracic level corresponding to maximal pain/dermatomal involvement, and was repeated every 48 hours for a total of three sessions.
  Arms: Ultrasound-guided thoracic paravertebral block (TPVB) with local anesthetic + corticosteroid

SUMMARY:
Background: Acute herpes zoster causes severe neuropathic pain and may progress to postherpetic neuralgia (PHN). This study aims to evaluate ultrasound-guided thoracic paravertebral block with local anesthetic and steroid in reducing acute pain and PHN incidence.

Methods: This prospective randomized study included 100 patients diagnosed with acute thoracic herpes zoster (rash ≤14 days, NRS ≥4). Participants were allocated into two groups: a control group receiving standard medical treatment and an intervention group receiving standard treatment in addition to an ultrasound-guided thoracic paravertebral block with (0.25% bupivacaine + 40 mg methylprednisolone) at 48-72-hour intervals. Pain intensity was assessed at baseline and during follow-up. The incidence of postherpetic neuralgia was recorded. Secondary outcomes included analgesic consumption and patient satisfaction.

ELIGIBILITY:
Eligibility Criteria Inclusion Criteria

Age 45-65 years

Diagnosed with acute thoracic herpes zoster

Rash duration ≤ 14 days

Moderate to severe pain, defined as NRS ≥ 4

Total sample size: 100 patients

Exclusion Criteria

Contraindications to thoracic paravertebral block, including:

Coagulopathy

Infection at the injection site

Allergy to local anesthetics or steroids

Immunosuppression or ongoing chemotherapy

Pre-existing chronic pain in the same affected region

Severe cognitive impairment or psychiatric illness preventing reliable pain assessment

Pregnancy or lactation

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2025-09-20 (Actual); Study Completion 2025-10-10 (Actual)

PRIMARY OUTCOMES:
The primary outcome was the incidence of postherpetic neuralgia (PHN), defined as a Numerical Rating Scale (NRS) pain score ≥4 persisting 90 days after rash onset. | till 3 month
  The primary outcome was the incidence of postherpetic neuralgia (PHN), defined as a Numerical Rating Scale (NRS) pain score ≥4 persisting 90 days after rash onset.

CONTACTS AND LOCATIONS:
Locations (1):
- Marwa Mahmoud Rady, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No
Plan Description
  De-identified individual participant data (IPD) will not be shared outside the study team.
  Access Criteria
  Not applicable.